CLINICAL TRIAL: NCT06788288
Title: The Long-term Impact of the Usage of New Generation Massage Chairs on Quality and Quantity of Sleep-in Individuals Suffering from Insomnia.
Brief Title: The Long-term Impact of Massage Chairs on Sleep Quality.
Acronym: autosleepilot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Collaborators: University of Nicosia (Other)
Responsible Party: Principal Investigator, Giorgos K. Sakkas, Associate Professor, University of Thessaly
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2334-5/4-2/7.2.2024
Record Dates: First submitted 2025-01-16; First posted 2025-01-23 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Insomnia
Keywords: poor sleepers; stress; fatigue
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Fatigue

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 - On-Off-On (Experimental): Participants will follow a crossover design with a one-month interval period for three months in total. Participants will be randomly assigned into two equal-sized groups receiving the intervention (massage) following a distinct pattern: for the Group-1: one month on, one month off, one month on. During the "on" period, the massage chair will be located at the participant's house while during the "off" period, the massage chair will be removed from the participant's house (washout period).
  Interventions: Other: Massage Chair session; Other: Washout period
- Group 2 - Off-On-Off (Experimental): Participants will follow a crossover design with a one-month interval period for three months in total. Participants will be randomly assigned into two equal-sized groups receiving the intervention (massage) following a distinct pattern: for the Group-2: one month off, one month on, one month off. During the "on" period, the massage chair will be located at the participant's house while during the "off" period, the massage chair will be removed from the participant's house (washout period).
  Interventions: Other: Massage Chair session; Other: Washout period

INTERVENTIONS:
Other: Massage Chair session — The intervention is composed of a full-body relaxation massage offered by an automatic electric massage chair. The intervention will last for 3 months while the participant will change between massage and washout periods.
  Other Names: Automatic Electric Massage chair
Other: Washout period — During this phase, participants will spend on month without any intervention (massage) accounting for a washout period.
  Other Names: no intervention

SUMMARY:
Modern technology is reshaping the massage industry, improving relaxation and well-being with pioneering devices. The automatic massage chairs stand as a testament to this evolution, integrating ergonomic design with advanced massage techniques to facilitate deep tissue relaxation, and sleep quality and enhance overall well-being.

Aim: The aim of the current study is to assess the long-term impact of the new generations of massage chairs prior to bed-time in aspects related to sleep and quality of life in individuals with severe symptoms of insomnia.

DETAILED DESCRIPTION:
Study Design The current study will assess the impact of daily usage (30 consecutive automatic massage sessions) of deep relaxation full body massage sessions using the 4D new generations' massage chairs in individuals suffering from insomnia. The massage chair will be located in patients' house/bedroom during the whole trial period.

Participants will follow a crossover design with one-month interval period for three months in total. Participants will be randomly assigned into two equal-sized groups receiving the intervention (massage) following a distinct pattern: for the Group-1: one month on, one month off, one month on, and for Group_2: one month off, one month on, one month off. During the "on" period, massage chair is located at participant's house while during the "off" period, massage chair is removed from participant's house.

During the "on" periods, participants could use the massage chair prior to bed time (last action before sleeping) and select from one of twelve programmed relaxation massage options. They were required to use the chair for at least 30 minutes daily, primarily before going to bed. The study was approved by the Human Research and Ethics Committee of the University of Thessaly (2334-5/4-2/7.2.2024). All Subjects gave their written informed consent prior to study participation.

Procedure All measurements will be conducted at the participants' own homes. Massage sessions will be performed in the participants' home prior to bedtime, utilizing the automatic massage chair provided during the study period.

The initial screening requires that all participants score ≥16 on the Athens Insomnia Scale (AIS-8). The Pittsburgh Sleep Quality Index (PSQI) was provided for participants to complete every 30 days over the three-month period. Additionally, during the first visit, all participants completed a series of validated questionnaires assessing quality of life, depression score, sleep quality, stress, and general fatigue. The same questionnaires were also completed during the final visit. After each visit and immediately after the completion of the 30 min automatic massage, participants will be connected to the portable polysomnography system and they will stay alone to follow their bedtime routine. The study recording will be completed when the participant wakes up and disconnects the system.

Questionnaires The following questionnaires will be administered using the interview method by experienced researchers.

* The Athens Insomnia Scale 1 and the Pittsburgh Sleep Quality Index (PSQI) will be used to assess sleep quality and the existence of any sleep abnormalities.
* The Short Form survey 36-item 36 quality of life questionnaire (SF-36) will be used to assess the health-related quality of life.
* The Beck Depression Inventory (BDI) questionnaire will be used for the assess symptoms of depression.
* The Perceived Stress Scale (PSS) will be used to assess the stress levels.

Body Composition Body composition will be assessed using anthropometric measurements, including BMI and bioelectrical impedance analysis with a Tanita DC-360S device (Tanita Corporation, Tokyo, Japan), following standard methodology.

Sleep Assessment A portable sleep monitoring system will be used to assess sleep quality and quantity (Home Sleep Test, Somnomedics, GmbH, Germany). The system records EEG, EOG, and EMG signals overnight. EEG data will be analyzed in 30-second epochs using SomnoMedics PSG analysis software (Domino panel ver. 3.0.0.8) with manual editing. The HomeSleepTest REM+ device will be used for PSG, with electrodes placed according to the 10/20 system on key brain regions: Fp1 (left) and M1 for EEG, and near the eyes for EOG. This setup ensures accurate monitoring of sleep architecture and high-fidelity recordings of brain activity and eye movements.

Analysis of the sleep study will be reported as follows: Total Sleep Time (total amount of sleep time scored during the total recording time); Sleep Efficiency (Total sleep time/Time in bed); Sustained Sleep Efficiency (Total sleep time/(Time in bed - Sleep laten-cy stage 2); Sleep Latency (the period of time it takes for a person to fall asleep after they have gone to bed and tried to initiate sleep); Sleep Latency N1 (the period of time between wakefulness and when sleep begins); Sleep Latency N2 (the period of time between time in bed and sleep onset stage 2); REM Latency (the amount of time elapsed between the onset of sleep to the first REM stage).

Massage Session Automatic Electric Massage Chair (AEMC) The Z1 Full Body 4D Massage Chair (Z1-SL Massage Chair, China, www.back2life.gr) will be used in the current study. The Z1-SL chair features a curved rail mechanism for both S-shaped (horizontal) and L-shaped (vertical) massages, covering areas from the head down toes. It includes 58 air cushions for air compression massage, while intelligent mechanical arms, rotating 360°, follow the body's contour, scanning and targeting specific areas for treatment.

The chair integrates a 4D massage system with professional techniques such as kneading, tapping, shiatsu, stretching, air compression, roller, and thermal massage. These techniques allow multidimensional effects in width, length, and depth, tailored to individual needs. Twelve automated programs vary in intensity, and the roller mechanism adjusts to body widths of 3 to 22 cm for focused application to areas like the cervical spine, back, and lower back.

The chair's infrared preheating function (carbon fiber-based) enhances relaxation and circulation by heating the back, pelvis, and thighs. This feature, combined with an extendable foot section and an airbag/roller system, ensures comfort for individuals of different sizes, providing muscle relaxation, fatigue relief, and improved blood circulation.

ELIGIBILITY:
Inclusion Criteria:

* score of ≥16 on the Athens Insomnia Scale (AIS-8)

Exclusion Criteria:

* history of mental illness,
* history of epilepsy
* acute or chronic condition that would limit the ability of the patient to participate in the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Sex at birth
Enrollment: 20 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Sleep Efficiency | At baseline, after each month and at the end of the 3 months period.
  Total sleep time over Time spend in bed
Insomnia Score | At baseline, after each month and at the end of the 3 months period.
  For the calculation of the Insomnia score, the Athens Insomnia Scale (AIS-8) will be used. The score ranges from 0 - 24 with a higher number implying worse insomnia symptoms.

SECONDARY OUTCOMES:
Sleep Quality Score | At baseline, after each month and at the end of the 3 months period.
  The Pittsburgh Sleep Quality Index (PSQI) will be used to assess sleep quality and the existence of any sleep abnormalities. The score ranges from 0 - 21 with a higher score implying worse sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Giorgos Sakkas, PhD, Study Chair — University of Thessaly
Locations (1):
- School of Physical Education, Sports and Dietetics, TEFAA, Trikala, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: Yes
When the data are available, we will provide a link to the data at the ClinicalTrials.gov record in the Available IPD/Information field in the References module of the Protocol Section.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: January 2026 - January 2027
Access Criteria: Written request

REFERENCES:
- [Background] Xie J, Fu M, Liu T, Li S, Liu G, Wang J, Ji C, Zhang T. Clinical studies on the electric automatic massage therapy for recovery of acute sports fatigue. Technol Health Care. 2023;31(S1):185-197. doi: 10.3233/THC-236016. PMID 37038791
- [Background] Kim JW, Lim AR, Lee JY, Lee JY, Lee S, Choi YJ, Kim YH, Park KH. The clinical effect of an electric massage chair on chemotherapy-induced nausea and vomiting in cancer patients: randomized phase II cross-over trial. BMC Complement Med Ther. 2024 Apr 19;24(1):163. doi: 10.1186/s12906-024-04464-8. PMID 38641782
- [Background] Khairudin MN, Vallikkannu N, Gan F, Hamdan M, Tan PC. Electric massage chairs reduce labor pain in nulliparous patients: a randomized crossover trial. Am J Obstet Gynecol MFM. 2024 Apr;6(4):101324. doi: 10.1016/j.ajogmf.2024.101324. Epub 2024 Mar 4. PMID 38447674